CLINICAL TRIAL: NCT06778512
Title: LcProt: Proteomics Longitudinal Cohort Study on Lung CancerProspective Longitudinal Cohort Study of Lung Cancer Based on Peripheral Blood and Tissue Proteomics
Brief Title: LcProt: Proteomics Longitudinal Cohort Study on Lung Cancer
Status: Recruiting | Type: Observational
Sponsor: The First Affiliated Hospital of Guangzhou Medical University (Other)
Responsible Party: Principal Investigator, Jianxing He, Professor, The First Affiliated Hospital of Guangzhou Medical University
Other Study IDs: LcProt; ES-2924-051-02 (Other: First Affiliated Hostipal of Guangzhou Medical University)
Record Dates: First submitted 2025-01-12; First posted 2025-01-16 (Actual); Last update posted 2025-01-16 (Actual); Status verified 2025-01

CONDITIONS: Lung; Lung Cancer; Cancer; NSCLC
Keywords: Lung cancer; Proteomics; Protein; NSCLC
MeSH Terms: conditions — Lung Neoplasms; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Using tissue and peripheral blood proteomics to distinguish the benign and malignant nature of lung cancer in patients, as well as to evaluate therapeutic efficacy and long-term prognosis during the t — Peripheral blood samples from enrolled participants will be drawn, or lesion tissues will be obtained through procedures such as biopsy or surgery, followed by quantitative proteomics analysis using mass spectrometry.
  Other Names: Draw peripheral blood; Obtain lesion tissue

SUMMARY:
This study will utilize tissue and peripheral blood samples for proteomics analysis and establish a longitudinal proteomics cohort at multiple critical treatment time points to explore the research value of proteomics in the diagnosis and treatment of lung cancer. The study includes key time points such as screening, postoperative efficacy prediction, and efficacy prediction after medication.

ELIGIBILITY:
Inclusion Criteria:

1. Signing of the informed consent form;
2. Male or female, aged 18-75 years;
3. Patients with lung nodules confirmed by CT examination;
4. Good preoperative pulmonary function cooperation and complete reporting;
5. Preoperative chest single/dual phase CT scans without significant artefacts and with complete imaging;
6. The interval between preoperative pulmonary function and single/dual phase CT scans does not exceed one month.

Exclusion Criteria:

1. Poor preoperative pulmonary function cooperation or missing reports;
2. Preoperative chest single/dual phase CT scans exhibit significant artefacts or image omission;
3. The interval between preoperative pulmonary function and single/dual phase CT scans exceeds one month;
4. Complication with severe respiratory disorders (such as lung transplantation, pneumothorax, giant bullae, etc.);
5. Coexisting with other severe functional impairments;
6. Patients with obstructive lesions such as airway or esophageal stenosis;

(8) Medication use before pulmonary function testing that does not meet the cessation guidelines; (9) Pulmonary function report quality graded D-F.

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with lung nodules confirmed by CT examination.
Sampling Method: Non-Probability Sample
Enrollment: 2500 (Estimated)
Dates: Start 2019-06-01 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Area Under the Curve | 3 years
  AUC, or Area Under the Curve, is a commonly used metric in statistical and machine learning models, particularly for evaluating the performance of classification models. It refers to the area under the Receiver Operating Characteristic (ROC) curve, which plots the true positive rate (sensitivity) against the false positive rate (1-specificity) at various threshold settings. An AUC value ranges from 0 to 1, where:
  * 1 indicates a perfect model,
  * 0.5 suggests a model no better than random guessing,
  * < 0.5 reflects a model performing worse than random.
  In clinical studies, AUC is often used to assess diagnostic tests, where a higher AUC indicates better test accuracy in distinguishing between conditions (e.g., disease vs. no disease).

SECONDARY OUTCOMES:
Differentially Expressed Proteins | 3 years
  Differential proteins, or differentially expressed proteins (DEPs), refer to proteins that show significant changes in expression levels between different biological or experimental conditions, such as disease vs. healthy states, treated vs. untreated groups, or across time points in longitudinal studies. These proteins are identified through quantitative proteomics techniques, including mass spectrometry or label-free methods, and analyzed using statistical or bioinformatics tools to determine significance.

CONTACTS AND LOCATIONS:
Locations (1):
- the First Affiliated of Guangzhou Medical University, Guangzhou, Guangdong, China